CLINICAL TRIAL: NCT01705756
Title: A Randomized Placebo-Controlled Study of the Efficacy and Safety of Kineret (Anakinra), in Adult Patients With Colchicine-Resistant Familial Mediterranean Fever
Brief Title: Kineret (Anakinra), in Adult Patients With Colchicine-Resistant Familial Mediterranean Fever
Acronym: FMF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof.Avi Livneh, Principal Investigator, Head of Internal Medicine "F" , Director of national center of FMF, Israel, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-11-8557-AL-CTIL
Record Dates: First submitted 2012-09-27; First posted 2012-10-12 (Estimated); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Familial Mediterranean Fever
Keywords: Colchicine; Anakinra; Colchicine resistance; Familial Mediterranean fever
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vehicle (Placebo Comparator): •Patients randomized to placebo will receive syringes identical to active drug (100 mg prefilled syringes for subcutaneous injection) filled with drug vehicle
  Interventions: Drug: Kineret
- Kineret (Anakinra) (Experimental): Patients randomized to active drug will receive Kineret (Anakinra), 100 mg prefilled syringes for subcutaneous injection, once a day for 4 months. The syringes will arrive relabeled from the supplier (SOBI) to Sheba Medical Center. They will be stored at the PI's store room in a temperature controlled refrigerator.
  Interventions: Drug: Kineret

INTERVENTIONS:
Drug: Kineret — Patients randomized to active drug will receive Kineret(Anakinra), 100 mg prefilled syringes for subcutaneous injection, once a day for 4 months. The syringes will arrive relabeled from the supplier (SOBI) to Sheba Medical Center. They will be stored at the PI's store room in a temperature controlled refrigerator.
  Other Names: Anakinra

SUMMARY:
FMF is the most common periodic fever with a worldwide patient population estimated as 150,000, mainly located in the Eastern Mediterranean basin. colchicine is the established therapy of choice ,however, around 20.000 patients worldwide fail to respond or cannot tolerate therapeutic doses, thereby suffering from recurrent debilitating, severe, painful attacks of peritonitis, pleuritis and synovitis and are at risk to die from reactive amyloidosis .Mutation-induced reduction in pyrin/ marenostrin activity is thought to underlie the disease by leading to NALP3 inflammasome activation ,and thereby to IL-1β related burst of inflammation.

The IL-1 receptor antagonist Kineret (Anakinra), seems to be the most appropriate response to the uncontrolled IL-1β elevation. Indeed, an increasing number of reports over the last few years indicate a good response to Kineret (Anakinra), in colchicine-resistant FMF ,also in children ,however, no controlled study has thoroughly evaluated the efficacy and safety of this treatment.

Study outline:

The study aims to run at the FMF centre in Sheba Medical Center, covering more than 10,000 patients. The study will evaluate the effect of recombinant IL-1 receptor antagonist, Kineret (Anakinra), on the frequency of FMF attacks in patients that, despite maximum tolerable dose of colchicine, present with more than one attack per month.

The study is designed as a randomised, placebo-controlled, double-blind study. 50 patients will be randomised to treatment with either Kineret (Anakinra), or placebo treatment for 4 months.

ELIGIBILITY:
Inclusion Criteria:

A subject must fulfil the following criteria in order to be included in the study:

1. FMF diagnosed as per the Tel-Hashomer criteria -(Criteria for the diagnosis of familial Mediterranean fever. Arthritis Rheum.1998 Aug; 41(8):1516-7-Livneh A, Langevitz P, Zemer D, Zaks N, Kees S, Lidar T, Migdal A, Padeh S, Pras M).
2. 18-65 years of age
3. Verified as mutations in both alleles of the MEFV gene, thus including homozygous and compound heterozygous patients
4. Patient compliant with maximum tolerable dose of colchicine (up to 3 mg/day)
5. At least one FMF attack per month in chest, abdomen or joints (definition of attack see above)
6. Adequate contraception for sexually active male and female patients

Exclusion Criteria:

The presence of any of the following will exclude a subject from inclusion in the study:

1. Patient pregnant at enrolment visit
2. Prior or existing malignancy
3. Active infection
4. Manifest renal failure with Creatinine clearance <30mL/min as determined by the equation Creatinine clearance (ml/min) = (140-age) x Wight (Kg) /72 x serum creatinine (mg/dcl) For women one should multiply the results by 0.8
5. Live vaccinations last three months before enrolment
6. Sociopsychological state threatening compliance with the treatment protocol
7. Alcohol or substance abuse
8. Concomitant medication with biological or anti-rheumatic disease-modifying drugs or systemic steroids
9. Any prior use of IL-1 inhibitory drugs
10. Associated disease that could interfere with clinical assessment:

    1. Rheumatic disorder
    2. Systemic disease, e.g. autoimmune or other autoinflammatory disorder, diabetes, hypertension, vasculitis, Behçet's disease
    3. Gastrointestinal disorder, e.g. Crohn's disease, ulcerative colitis, irritable bowel syndrome
    4. Cardiovascular disorder, e.g. post myocardial infarction, angina
    5. Pulmonary disorder, e.g. COPD, pulmonary hypertension
    6. Any other condition which in the opinion of the investigator makes the subject unsuitable for inclusion
11. Enrolment in another concurrent clinical study, or intake of an investigational drug, within three months prior to inclusion in this study
12. Failure or refusal to cooperate with given instructions

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with less than a mean of one FMF attack per month | 4 months
  Total number of FMF attacks in abdominal, thoracic, skin or joint locations during the observational period (4 months) as recorded in the patient diary, devided by 4 for each patient will result in number of attacks per one month. The number of patients with less than 1 attack per month will be compared between the 2 study groups

SECONDARY OUTCOMES:
Number of serious adverse events | 4 months
  Secondary endpoint is defined as total number of serious adverse events per 4 months in each study group. SAE is defined as an adverse event that meets one or more of the following criteria/outcomes:
  * Death
  * Life-threatening (i.e., at immediate risk of death)
  * In-patient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect

CONTACTS AND LOCATIONS:
Overall Officials: Avi Livneh, professor, Principal Investigator — Sheba Medical Center, Tel- Hashomer, Ramat- Gan, Israel.
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Derived] Ben-Zvi I, Kukuy O, Giat E, Pras E, Feld O, Kivity S, Perski O, Bornstein G, Grossman C, Harari G, Lidar M, Livneh A. Anakinra for Colchicine-Resistant Familial Mediterranean Fever: A Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2017 Apr;69(4):854-862. doi: 10.1002/art.39995. PMID 27860460